CLINICAL TRIAL: NCT01614080
Title: Outcome of Patients Treated by iv Rt-PA for Cerebral Ischaemia According to the Ratio Sc-tPA/Tc-tPA in the Administered Rt-PA
Brief Title: Outcome of Patients Treated by iv Rt-PA for Cerebral Ischaemia According to the Ratio Sc-tPA/Tc-tPA
Acronym: OPHELIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 10.677; 2010_04 (Other: sponsor)
Record Dates: First submitted 2012-04-23; First posted 2012-06-07 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Stroke, Acute; Drug Toxicity
Keywords: Stroke; Ischemic stroke; thrombolysis; toxicity of t-PA
MeSH Terms: conditions — Stroke; Drug-Related Side Effects and Adverse Reactions; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High sc-tPA/tc-tPA ratio group: A threshold value of the sc-tPA/tc-tPA ratio will be defined as the median value found in the population. The High sc-tPA/tc-tPA ratio group will be defined as the group of patients with a sc-tPA/tc-tPA ratio higher than the median
- Low sc-tPA/tc-tPA ratio: A threshold value of the sc-tPA/tc-tPA ratio will be defined as the median value found in the population. The Low sc-tPA/tc-tPA ratio group will be defined as the group of patients with a sc-tPA/tc-tPA ratio lower than the median

SUMMARY:
intravenous rt-PA is effective to reduce the risk of death or dependency after ischaemic stroke. This effect is due to an early recanalization secondary to the lysis of the clot. However this effect may be counterbalanced by the increased risk of bleeding and also the neurotoxicity of rt-PA, which has been shown in animals to depend on the ratio single chain (sc) / double chain (tc) in the rt-PA administered. The main objective of OPHELIE is to determine whether the functional outcome after treatment by iv rt-PA depends on the ratio sc-rtPA / tc-rtPA. Secondary objectives were to identify the influence on the risk of brain haemorrhage, and the influence of the cognitive state (OPHELIE-COG substudy).

DETAILED DESCRIPTION:
OPHELIE is a multicenter study conducted in France in 25 centers where patients treated by iv rt-PA will be included. Patients are treated according to the local protocol, without any modification specifically for this study. A sample of 2 drops of the rt-PA used for the treatment is stored for analysis, to determine the sc-tPA/tc-tPA ration (immunostaining).

700 patients are needed for the study assuming that a difference of 5% will be found in the primary outcome measure (modified Rankin scale 0-1 at 3 months) with alpha and beta risks respectively of 5% and 20%.

The participating clinical centres recruit altogether more than 500 patients per year for thrombolysis. Assuming that 70% will be eligible, the recruitment should take less than 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Being treated by iv tPA for acute cerebral ischaemia

Exclusion Criteria:

* absence of reliable informant
* no rtPA left in the syringe after treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in routine by iv t-PA for acute ischaemic stroke
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
OPHELIE | Month 3
  The proportion of the patients with modified Rankin Scale 0-1

SECONDARY OUTCOMES:
OPHELIE | 7 days
  The proportion of the patients with symptomatic intra cerebral haemorrhage according to ECASS 2 definition

CONTACTS AND LOCATIONS:
Overall Officials: Kei MURAO, MD, Study Director — University Lille 2; Denis VIVIEN, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Didier LEYS, MD, PhD, Principal Investigator — Lille University Hospital
Locations (1):
- Lille University Hospital, Lille, France

REFERENCES:
- [Derived] Caparros F, Kuchcinski G, Drelon A, Casolla B, Moulin S, Dequatre-Ponchelle N, Henon H, Cordonnier C, Pruvo JP, Leys D. Use of MRI to predict symptomatic haemorrhagic transformation after thrombolysis for cerebral ischaemia. J Neurol Neurosurg Psychiatry. 2020 Apr;91(4):402-410. doi: 10.1136/jnnp-2019-321904. Epub 2020 Feb 3. PMID 32015090
- [Derived] Leys D, Hommet Y, Jacquet C, Moulin S, Sibon I, Mas JL, Moulin T, Giroud M, Sagnier S, Cordonnier C, Medeiros de Bustos E, Turc G, Ronziere T, Bejot Y, Detante O, Ouk T, Mendyk AM, Favrole P, Zuber M, Triquenot-Bagan A, Ozkul-Wermester O, Montoro FM, Lamy C, Faivre A, Lebouvier L, Potey C, Poli M, Henon H, Renou P, Dequatre-Ponchelle N, Bodenant M, Debruxelles S, Rossi C, Bordet R, Vivien D; OPHELIE investigators and the STROKAVENIR network. Proportion of single-chain recombinant tissue plasminogen activator and outcome after stroke. Neurology. 2016 Dec 6;87(23):2416-2426. doi: 10.1212/WNL.0000000000003399. Epub 2016 Nov 4. PMID 27815401